CLINICAL TRIAL: NCT02159781
Title: Effect of Periodontal Treatment on Salivary Biomarkers.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, Eran Front, Unit of Periodontology - Department of Oral and Maxillofacial surgery, The Baruch Padeh Medical Center, Poriya
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-1476.CTIL
Record Dates: First submitted 2014-05-28; First posted 2014-06-10 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- periodontal treatmnent (Experimental)
  Interventions: Procedure: periodontal treatment - scaling and root planning

INTERVENTIONS:
Procedure: periodontal treatment - scaling and root planning

SUMMARY:
The investigators plan to recruit 40 healthy patients referred to the unit of Periodontology, diagnosed with generalized moderate - severe chronic periodontitis.

treatment will include 4 - 6 sessions of scaling + root planning, oral hygiene instructions and motivation.

Whole saliva will be collected at intake and 8 - 14 weeks post periodontal treatment.

Saliva will be analyzed for trans locator protein. Study hypothesis: Periodontal treatment has an affect on saliva components.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients
* moderate - sever chronic periodontitis

Exclusion Criteria:

* systemic disease
* pregnancy
* subjects under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Whole saliva & translocator protein (TSPO) | Intake of patients than 8 - 12 weeks after periodontal treatment (scaling & root planning)
  Change in whole saliva & translocator protein (TSPO) post periodontal treatment

SECONDARY OUTCOMES:
Periodontal measurements (periodontal pocket depth, bleeding on probing & clinical attachment level) | Intake 8 - 12 weeks post periodontal treatment (scaling & root planning)
  periodontal probing depth, bleeding on probing and clinical attachment level.